CLINICAL TRIAL: NCT04504058
Title: Construction of Nutritional Optimization Path for Prevention and Treatment of Common Mental Diseases Based on Skin Response Quantification Instrument
Brief Title: Construction of Nutritional Path for Mental Diseases
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Principal Investigator, Tianhong ZHANG, Associate Professor, Shanghai Mental Health Center
Other Study IDs: 2020080501
Record Dates: First submitted 2020-08-05; First posted 2020-08-07 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Clinical High-risk
Keywords: nicotinic acid; skin flush reaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — fingertip blood fat spectrum detection
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- UFACH: Unsaturated Fatty Acid in Clinical High-risk
  Interventions: Other: routine clinical treatment

INTERVENTIONS:
Other: routine clinical treatment — Participants will be informed that this is not a treatment study and it involves naturalistic follow-up without any extra intervention. They will otherwise follow the routine clinical treatment procedure.

SUMMARY:
The project will focus on the major technical difficulty of "lack of effective nutritional intervention measures for early risk of common mental diseases in China", and rely on the platform of psychiatric risk identification and treatment specialty of Shanghai Mental Health Center, an authoritative institution in the field of mental health, and focus on the effective application of the domestic independent research and development of the artificial intelligence nicotinic acid skin flushing reaction quantification instrument.

DETAILED DESCRIPTION:
Based on the biological data of one of the world's largest cohort of psychiatric patients with early phase and risk, nicotinic acid reaction pictures were introduced as biological information for the first time in nutritional intervention of psychiatric risk prevention and control.

Exploration of machine learning and big data analysis methods, based on the objective quantitative evaluation tool, combined with fingertip blood fat spectrum detection, to construct the optimization scheme and targeted non drug intervention measures of nutritional supplement for common mental diseases.

From the perspective of antioxidant stress and nutritional supplement, a new clinical pathway for the prevention and treatment of mental diseases with artificial intelligence products as screening, early warning and guidance prevention will be established.

ELIGIBILITY:
Inclusion Criteria:

* be aged 14 to 45-year-old；
* have had at least 6-years of primary education；
* be drug-naïve；
* be understanding the survey, be willing to enrol in the study and sign the informed consent；
* Through the Structured Interview for Prodromal Syndromes/Scale of Prodromal Symptoms (SIPS/SOPS), the participants should meet the Criteria of Prodromal Syndrome. Participants should fulfil at least one of the prodromal syndrome criteria: (1) brief intermittent psychotic syndrome, (2) attenuated positive symptom syndrome, or (3) genetic risk and deterioration syndrome.

Exclusion Criteria:

* Through the Mini-International Neuropsychiatric Interview (MINI), Axis I mental disorders such as schizophrenia, affective disorders, and anxiety spectrum disorders will be excluded;
* Acute or chronic renal failure; liver cirrhosis or active liver diseases;
* Abnormal laboratory tests results judged by the researchers to be clinically significant and considered to affect the efficacy of the test drugs or the safety of the subjects;
* Severe or unstable physical diseases, including: neurological disorders (delirium, dementia, stroke, epilepsy, migraine, etc.), congestive heart failure, angina pectoris, myocardial infarction, arrhythmia, hypertension (including untreated or uncontrolled hypertension), malignant tumours, immune compromise, and blood glucose above 12 mmol/L;
* Alcohol abuse within 30 days, or alcohol or drug dependence within 6 months before the trial;
* Pregnant or lactating women, or women in childbearing age who are positive in urine human chorionic gonadotropin test, or men and women who do not take effective contraceptive measures or plan for pregnancy within 3 months after the initiation of the trial;
* Stroke within the last month;
* Participating in any clinical trial within 30 days before the baseline;
* Other situations judged by the investigators not to be suitable for the clinical trial.

Ages: 14 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Help-seeking first-visit participants will be consecutively recruited from the Shanghai Psychotherapy and Psychological Counselling Centre at the Shanghai Mental Health Centre. They will be screened for eligibility by their clinicians.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-10-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Conversion to psychosis | 4 weeks
  It will be determined using the criteria for the Presence of Psychotic Symptoms from SIPS. Specifically, the conversion will be defined by the presence of level 6 positive symptoms (the rating "6" refers to severe and psychotic symptoms) identified as either dangerous, disorganised, or occurring at least one hour a day on average, over four days a week for at least 16 hours.
Poor function | 4 weeks
  It will be determined by GAF score. Specifically, poor function outcome is defined as the GAF score of less than 60 at the follow-up point.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Mental Health Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code